CLINICAL TRIAL: NCT06828510
Title: Evaluation of the ORTHOPUS Partner Arm in People With Disabilities Needing for Robotic Assistance to Compensate for Upper Limb Deficiency
Brief Title: Evaluation of ORTHOPUS Partner Arm in People With Disabilities Needing for Robotic Assistance to Compensate for Upper Limb Deficiency
Acronym: MS PARTNER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP241006; 2024-A02447-40 (Registry Identifier: IDRCB)
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Disability Physical
Keywords: disability; robotic; impairment; upper limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ORTHOPUS PARTNER (Experimental)
  Interventions: Device: With device

INTERVENTIONS:
Device: With device — Medical Device Installation Visit (V2, Day 0 + 21 ± 10 days): This visit, lasting approximately 1.5 hours, takes place in a consultation room at the center. A representative from ORTHOPUS adapts and installs the Partner on the patient's wheelchair, and an initial training session on the use of the medical device is provided.
  Use of the Medical Device in Ecological Conditions (between V2 and V3): Between Day 21 and Day 42, the patient is invited to use the MD without restrictions in real-life conditions.
  Final Evaluation Visit (V3, three weeks after V2, up to four weeks if necessary): The assessment session for the primary outcome-functional goal achievement using the GAS method-is conducted following the SCED (Single-Case Experimental Design) procedure, with multiple introduction-withdrawal phases and randomized phase sequencing and repeated measures :

SUMMARY:
The study is a prospective, multicenter, interventional, open clinical trial, in Single Case Experimental Design (SCED) in multiple introduction withdrawal, controlled, randomized.

DETAILED DESCRIPTION:
The function of the upper limb associated with gripping is essential for carrying out activities of daily living (ADL): personal care, productive activities, leisure, etc. The upper limbs therefore have not only a functional dimension (bringing together, moving away, holding, taking, bringing to the mouth, scratching, etc.) but also a social and anthropological one. As such, a limitation of functionality of the upper limb will have a very significant impact on the quality of life, independence, autonomy and participation of the subjects. When the impairment of a function is irreversible, rehabilitation care may involve the use of aids that either optimize or replace the function. Thus, the orthoses or devices used can either assist the movement if a minimum of muscular strength and control is still present, or completely replace the function if the functional deficit is complete. Using the proprietary robotic actuator, ORTHOPUS has developed the Partner for people with disabilities, with residual strength in the arm. This device is therefore intended for people with a loss of function in the upper limbs. It supports the mobility of the arm by anti-gravity compensation and must help to regain autonomy during ADLs. The Partner is CE marked and classified as a class 1 MD. The hypothesis of the Clinical Investigation is that the Partner medical device is effective in improving the functional capacities of the equipped upper limb (LM), in patients, children and adults, eligible for a robotic compensation Upper Limb Technical Aid, after a period of use of said technical aid in ecological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Have a loss of mobility in the upper limb (UL).
* Have minimal functional capacities in the upper limb, defined by a score between 1 and 4 on the Lovett scale for all muscle groups of the arm, except for the hand and wrist.
* Demonstrate effective distal motor skills in the upper limb to be fitted.
* Be an informed patient who has provided signed consent, or in the case of minors, have given assent along with the signed consent of legal guardians.
* A relative must be available for the installation visit, and either the patient or the relative must have the necessary equipment to record videos in ecological conditions (smartphone or tablet).)

Exclusion Criteria:

* Patients with cognitive or behavioral dysfunctions that may compromise adherence to instructions and procedures required for the trial (at the discretion of the investigator clinician).
* Patients already enrolled in an interventional clinical trial.
* History of fractures in the upper limb to be fitted within the six months preceding the inclusion visit in the trial.
* Any conditions or injuries that may interfere with functional assessments.
* Patients under legal guardianship or curatorship.
* Lack of health insurance coverage.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Personalized functional goal achievement score | Day 45
  Personalized functional goal achievement score, defined using the Goal Attainment Scaling (GAS) method, assessed after three weeks of Partner use, both with and without the Partner.
  The Goal Attainment Scale (GAS) is an individualized outcome measure involving goal selection and goal scaling that is standardized in order to calculated the extent to which a patient's goals are met.

CONTACTS AND LOCATIONS:
Overall Officials: Thibaud LANSAMAN, MD, Principal Investigator — SMR DEPARTMENT, Raymon Pincaré Hospital - APHP; Samuel POUPLIN, PhD, Study Director — PFNT DEPARTMENT, Raymon Pincaré Hospital - APHP

IPD SHARING:
Plan to Share IPD: Undecided